CLINICAL TRIAL: NCT06943378
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose and Dose Expansion Study to Assess the Safety, Tolerability and Pharmacokinetics of a Monoclonal Antibody, JST-010, in Healthy Adults
Brief Title: Ph1, Randomized, Double-Blind and Controlled, Dose Escalation and Expansion Study to Assess the Safety and Pharmacokinetics of JST-010 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Just-Evotec Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DDF3-CL101; MCDC No. W15QKN-16-9-1002 (Other: US Department of Defense)
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Pre-exposure Prophylaxis Against Pneumonic Plague in Healthy Adults
Keywords: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blinded, Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor and CRO
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- JST-010: The active investigational product (Active Comparator)
  Interventions: Biological: Monoclonal antibody JST-010
- JST-012 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Monoclonal antibody JST-010 — Active study drug
  Arms: JST-010: The active investigational product
Drug: Placebo — Placebo
  Arms: JST-012 Placebo

SUMMARY:
The goal of this clinical trial is to learn if a single dose of the study drug, JST-010, is safe and tolerable when administered by injection into the arm or thigh muscle of healthy men and women aged 18 to 55. The main questions it aims to answer are:

* Is a single injection of JST-010 safe?
* What is the concentration of the JST-01 in the blood over time?
* Do antibodies to JST-010 develop following a dose of JST-010?

Researchers will compare JST-010 to Placebo to see if there are any differences in the safety and tolerability of a single dose at different dose levels.

Participants will be confined to the clinic for the first 3 days. They will receive an injection on the second day, and then return for 9 more visits over the period of 1 year for:

* Physical exam with vital signs
* Electro-cardiogram (ECG)
* Bood collection for clinical labs and research samples
* Urine sample
* Assessment of potential adverse effects and medications taken

DETAILED DESCRIPTION:
This is a two-part, Phase 1, first-in-human (FIH), randomized, double-blind, placebo-controlled, single ascending dose (SAD) (Part 1) and dose expansion (Part 2) study to assess the safety, tolerability, and PK of a single dose of JST-010 administered IM to healthy participants.

Part 1 will comprise a minimum of 3 SAD cohorts (Cohorts A, B, and C, with 14 participants per cohort), each evaluating a single dose of JST-010 administered IM. In each SAD cohort, 2 sentinel participants will be randomized 1:1 such that one participant receives JST-010 and 1 participant receives placebo. Following a favorable blinded safety review committee (SRC) review of sentinel safety data collected through Day 8, the remainder of the cohort (12 non-sentinel participants) will be randomized 5:1 to JST-010 or placebo, and the first block of 6 participants (5:1 JST-010 to placebo) will be dosed. The SRC will review the safety data collected during the first 48 hours after dosing for the first block of 6 participants dosed to determine whether the second block of 6 participants can be dosed.

All safety data for all participants in the current cohort through Day 8 with cumulative prior safety data will be reviewed by the SRC in a blinded fashion for each dose cohort before escalating to the next dose cohort (for escalation from Cohort A to Cohort B and escalation from Cohort B to Cohort C); the SRC will have the ability to consult with the independent data monitoring committee (IDMC) as needed regarding these decisions. A recommendation on whether to implement Cohort D (along with a recommended dose of JST-010 to be evaluated in Cohort D) may be provided by the SRC following review of blinded safety data from Cohorts A, B, and C, or may be provided by the IDMC following review of unblinded safety, PK, and antidrug antibody (ADA) data from Cohorts A, B, and C.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women 18 to 55 years of age
2. BMI between 18 and 32 kg/m2
3. Negative serum pregnancy test
4. Use of highly effective birth control method(s) for a minimum of 60 days prior to consent and is willing to continue use for at least 12 months, or abstinence
5. In good general health as determined by medical history, exams and tests

Exclusion Criteria:

1. Acute illness or fever (≥100.4°F) within 7 days prior to dosing
2. Any history of receiving treatment, vaccine, or monoclonal antibodies (mAbs) against the Yersinia pestis bacterium
3. Receipt of any vaccine within 30 days prior to Screening, planned receipt of any vaccine prior to Day 1, or planned receipt of any vaccines before 45 days post-injection.
4. Any medical condition for which IM injections would be contraindicated in the opinion of the investigator (eg, bleeding disorders, anticoagulant therapy, and severe thrombocytopenia)
5. History of congenital or acquired immunodeficiency syndrome
6. Prior solid organ or bone marrow transplant
7. Use of systemic steroids, immunosuppressive agents, anticoagulants, or antiarrhythmics within 1 year prior. A single short course (ie, less than 14 days) is allowed provided it is concluded more than 6 months prior to Screening
8. Upper arm is with insufficient muscular tissue for IM injections or is obscured by tattoos or rash that may preclude accurate assessment of injection site reactions
9. Use of any medications started within 30 days prior to Day -1, including prescription medications, nutritional supplements, and over-the-counter medications

   * Vitamin supplements are allowed
   * Recommended doses of acetaminophen are allowed, except for 24 hours prior to dosing
   * Recommended doses of non-steroidal anti-inflammatory drugs (NSAIDs) (eg, aspirin, ibuprofen) are also allowed, except for 7 days prior to dosing
10. Positive human immunodeficiency virus (HIV-1/-2) antibody result by history or at Screening
11. Positive hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C antibody
12. Positive urine drug test or cotinine (indicating active current smoking) at Screening or Day -1, positive alcohol breath test at Screening or on Day -1, or suspected/known drug abuse and/or alcohol use disorder
13. Smoking or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 3 months before study drug dosing
14. Dosing in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer) of receiving the investigational drug prior to Screening
15. Progressive, unstable, or uncontrolled medical conditions that have required medical attention or changes to medication for medical reasons within 90 days prior to consent
16. History of allergic reactions or hypersensitivity reactions to other therapeutic antibodies or immunoglobulins
17. Receipt of any mAbs in the 12 months prior to Screening
18. High blood pressure
19. History of hyperprolinemia
20. Women who are either pregnant or breast-feeding
21. Vulnerable individuals (eg, military recruits, persons in compulsory detention, those with limited legal capacity)
22. Receipt of immunoglobulins or any blood products within 90 days prior to consent or planned receipt during the study period
23. Donation or loss of >500 mL of blood within 30 days or plasma within 7 days of Day 1; any planned donation of blood or plasma during the study period
24. History of any malignant neoplasm within the last 5 years, with the exception of adequately treated localized or in situ non-melanoma carcinoma of the skin or the cervix
25. Strenuous activity or contact sports within 48 hours before study drug dosing and through Day 8
26. History of relevant drug and/or food allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of a single dose of JST-010 when administered intramuscularly (IM) in healthy adults | 1) Local and systemic solicited AES from injection to Day 7, 2) All AEs post-injection to final visit at Week 48, 3) SAEs, MAAEs, and AESIs post-injection to final visit at Week 48
  1. Incidence of solicited local (injection site) and systemic AEs post-injection through Day 7 (with the inpatient and outpatient participant diaries being collected on Day 3 and Day 8, respectively).
  2. Incidence of unsolicited AEs through end of study (EOS).
  3. Incidence of SAEs, medically attended AEs (MAAEs), and AEs of special interest (AESIs) post-injection through EOS.

SECONDARY OUTCOMES:
Pharmacokinetic Cmax of JST-010 | From enrollment to the end of study at 48 weeks
  Maximum observed concentration (Cmax)
Pharmacokinetic Tmax of JST-010 | From enrollment to the end of study at 48 weeks
  Time to reach maximum observed concentration (Tmax)
Pharmacokinetic Tlast of JST-010 | From enrollment to the end of study at 48 weeks
  The timepoint with the last quantifiable concentration (Tlast)
Pharmacokinetic AUC0-D85 of JST-010 | From enrollment to the end of study at 48 weeks
  Area under the concentration versus time curve (AUC) from time 0 to Day 85 (AUC0-D85)
Pharmacokinetic AUC0-t of JST-010 | From enrollment to the end of study at 48 weeks
  Area under the concentration versus time curve (AUC) from time 0 to the timepoint with the last quantifiable concentration (AUC0-t)
Pharmacokinetic AUC0-inf of JST-010 | From enrollment to the end of study at 48 weeks
  AUC from time 0 extrapolated to infinity (AUC0-inf)
Pharmacokinetic t1/2 of JST-010 | From enrollment to the end of study at 48 weeks
  Terminal elimination half-life (t1/2)
Pharmacokinetic CL/F of JST-010 | From enrollment to the end of study at 48 weeks
  Apparent clearance after IM administration (CL/F)
Pharmacokinetic Vz/F of JST-010 | From enrollment to the end of study at 48 weeks
  Apparent volume of distribution after IM administration (Vz/F)
Evaluation of anti-JST-010 drug antibodies following IM administration of a single dose of JST-010 | From enrollment to the end of study at 48 weeks.
  Immunogenicity: ADAs that develop to JST-010 or are pre-existing prior to administration of JST-010 may be associated with potential allergic reactions and could negatively impact the effectiveness of JST-010. ADAs will be evaluated throughout the duration of the trial. Participants who develop any AE associated with the development of ADAs will be followed until such AEs are resolved, stable, or judged by the investigator to be not clinically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Las Vegas Clinical Research Unit, Las Vegas, Nevada, United States